CLINICAL TRIAL: NCT05472181
Title: The Effects of Brain Stimulation on Enhancement of Speech Fluency in Adults Who Stutter
Brief Title: The Effects of Brain Stimulation on Speech Fluency in Adults Who Stutter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS_stuttering
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Stuttering, Adult
Keywords: TMS; Stuttering; Supplementary Motor Area (SMA)
MeSH Terms: conditions — Stuttering | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a double-blinded between- and within-subjects crossover sham-controlled design across two different treatment phases to enhance the effects of behavioural training on stuttering.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Repetitive TMS) (Active Comparator): The rTMS group will receive 30 minutes of excitatory rTMS (i.e., 60 trains of 10 Hz pulses for 5 second with over 120% of motor threshold) over SMA combined with speech training (for 25 seconds during the 60 inter-train intervals) for five sessions
  Interventions: Device: rTMS (Repetitive TMS); Behavioral: Speech training
- Sham (Sham Comparator): The sham group will receive 30 minutes of sham rTMS (no magnetic stimulation) over SMA combined with speech training (for 25 seconds during the 60 inter-train intervals) for five sessions.
  Interventions: Behavioral: Speech training

INTERVENTIONS:
Device: rTMS (Repetitive TMS) — TMS stimulation produce electromagnetic pulses that can directly changes the neural firing in the brain. The rTMS applies the magnetic pulses in a repetitive manner, and can induce either an inhibitory or excitatory effect on cortical neurons. In this study we use high frequency rTMS (10 Hz) to provide the excitatory effect.
  Arms: rTMS (Repetitive TMS)
Behavioral: Speech training — The behavioural training will include reading sentences in which a syllable is spoken in time to a rhythmic beat.

SUMMARY:
The project is leading to investigate the effects of neuromodulation techniques on speech fluency among adults who stutter (AWS). While stuttering is responsive to a variety of treatments in childhood, this is not the case for AWS. Behavioural treatments to reduce stuttering for adults typically consist of speech restructuring methods, which involves the person using one of the altered speech patterns known to increase fluency, such as chorus reading, speaking in rhythm, and prolonging (smoothing/stretching out) speech sounds. Research has shown that behavioural interventions such as these change brain activation patterns in the regions associated with stuttering. Unfortunately, around 70% of AWS who receive these speech restructuring treatments do not maintain the benefits in the longer term and frequently re-present to speech clinics. The aim of this proposed research is to explore whether the brain stimulation using repetitive transcranial magnetic stimulation (rTMS) can consistently enhance effects of behavioural stuttering therapy by examining their responsiveness to the treatment across different outcome measures including a) immediate effect on different speaking contexts, and b) the maintenance of effects over one week after therapy.

ELIGIBILITY:
Inclusion Criteria:

- adults who stutter without any other speech, language or cognitive problems

Exclusion Criteria:

* have any history of neurological and other speech and language problems
* condition that are violating the safety criteria for TMS
* any history of epilepsy, and brain damage,
* having any metal plant or cardiac pace-maker in the body,
* current pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Stuttering severity | Immediately and one week after the treatment block
  The stuttering severity will be measured by Stuttering severity instrument-4 (SSI-4)

SECONDARY OUTCOMES:
Treatment satisfaction | one week after the treatment block
  For the assessment of subject satisfaction regarding the treatment, the following two Likert-type survey questions will be asked at weeks 1 post-treatment, to which the participants will respond: (1) How much do you think the treatment helped you to speak more fluently? (1 = not at all, 2 = a little, 3 = somewhat, 4 = a lot, 5 = totally); and (2) How often/much do you think the treatment helped you to feel less stressed in your communication? (1 = never or not at all, 2 = rarely or a little, 3 = sometimes or somewhat, 4 = often or a lot, 5 = always or totally).

CONTACTS AND LOCATIONS:
Locations (1):
- TMS Lab, Faculty of Education, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Bakhtiar M, Yeung TWY, Choi A. The application of neuronavigated rTMS of the supplementary motor area and rhythmic speech training for stuttering intervention. Int J Lang Commun Disord. 2024 Sep-Oct;59(5):1893-1905. doi: 10.1111/1460-6984.13039. Epub 2024 May 6. PMID 38711376